CLINICAL TRIAL: NCT00602290
Title: The Use of Methylphenidate to Improve Clinical Outcomes in Geriatric Depression: A Double-blind Placebo-Controlled Trial of Methylphenidate (Ritalin) Augmentation of Citalopram (Celexa) in Depressed Elderly Patients
Brief Title: Effectiveness of Methylphenidate in Improving Cognition and Function in Older Adults With Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Helen Lavretsky, MD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH077650 (NIH); R01MH077650 (NIH); DATR A4-GPX
Record Dates: First submitted 2008-01-23; First posted 2008-01-28 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2017-12

CONDITIONS: Depression
Keywords: Major Depression; Geriatric Major Unipolar Depression; Executive Cognitive Dysfunction; Elderly; Geriatric; Executive Cognitive Impairment; Quality of Life; Disability; Comorbidity; Medical Burden; Safety; Candidate Genes
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Citalopram; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 - Citalopram and placebo (Active Comparator): Participants will take a combination of citalopram and placebo for 16 weeks
  Interventions: Drug: Citalopram; Drug: Placebo
- 2 - Methylphenidate and placebo (Active Comparator): Participants will take a combination of methylphenidate and placebo for 16 weeks
  Interventions: Drug: Methylphenidate (MPH); Drug: Placebo
- 3 - Methylphenidate and Citalopram (Active Comparator): Participants will take a combination of methylphenidate and citalopram for 16 weeks
  Interventions: Drug: Citalopram; Drug: Methylphenidate (MPH)

INTERVENTIONS:
Drug: Citalopram — Citalopram dosage will be 20 to 60 mg a day prior to FDA warning limiting it to 20-40 mg in 2011. Participants will begin taking one 20-mg capsule once per day for 4 weeks, and this dosage may be increased or decreased depending on the participant's response to the medication or side-effect profile. Participants will continue on their assigned dosage of citalopram that will be titrated up after week 4 if clinical global impressions (CGI) scores were > 2 until treatment completion.
  Other Names: Celexa
  Arms: 1 - Citalopram and placebo; 3 - Methylphenidate and Citalopram
Drug: Methylphenidate (MPH) — MPH dosage will be 5 to 40 mg a day. Participants will initially take 1 capsule (2.5 mg) twice per day, which will be increased to a maximum up to 8 x 2.5 mg capsules twice per day. After Visit 11, MPH dosage will be gradually reduced over 2 weeks until participants are no longer taking any capsules.
  Other Names: Ritalin
  Arms: 2 - Methylphenidate and placebo; 3 - Methylphenidate and Citalopram
Drug: Placebo — Placebo pills will be taken in combination with the active pills. Participants will initially take 1 capsule twice per day, which will be increased to a maximum of 16 capsules twice per day matching methylphenidate, and 1-3 capsules matching citalopram. After Visit 11, placebo dosage will be gradually reduced over 2 weeks until participants are no longer taking any capsules.
  Arms: 1 - Citalopram and placebo; 2 - Methylphenidate and placebo

SUMMARY:
This study will evaluate the safety and effectiveness of methylphenidate in improving cognition and function in older adults with depression.

DETAILED DESCRIPTION:
Less than 50% of older adults with depression achieve remission and functional recovery in response to first-line antidepressant treatment. Most are left with significant residual symptoms, putting them at risk for illness relapse, frailty, and suicide. Improved understanding of the neurobiology of depression in older adults and mechanisms of treatment response may lead to better clinical management of depression. Methylphenidate (MPH) has long been used in the elderly and the medically ill to provide rapid improvement in depression, apathy, and fatigue. However, its potential beneficial effects on cognitive and functional outcomes in older adults with depression have not been studied. Combining MPH with the serotonergic antidepressant citalopram may result in better clinical outcomes than would using citalopram alone. This study will compare the safety and effectiveness of MPH combined with citalopram, MPH combined with placebo, and citalopram combined with placebo in improving thinking, memory, and speed of recovery in older adults with depression. The study will also evaluate selected dopamine- and serotonin-related gene relationships with mood, cognitive symptoms, and treatment response to MPH and citalopram.

Participation in this double-blind study will last 16 weeks. All potential participants will initially undergo comprehensive medical, neuropsychiatric, and cognitive assessments and genetic testing. These initial assessments will include questionnaires about depressive symptoms, a medical history, an electrocardiogram (ECG), and a blood draw for the genetic testing. Eligible participants will then be randomly assigned to one of three groups: MPH and citalopram, MPH and placebo, or citalopram and placebo. All participants will receive 16 weeks of treatment with their assigned medications. Study visits will occur weekly for the first 6 weeks of treatment and bi-weekly for the remainder of the study. During study visits, participants will undergo vital sign and weight measurements, answer questionnaires, and report any medication side effects. Blood will again be drawn at Visits 4 and 10, and the ECG will be repeated at Visit 10 if any cardiac symptoms occur. Most initial assessments will be repeated on Visit 13, the last study visit. Participants will also be contacted weekly by phone throughout the study to answer questions on how they are feeling and any possible side effects.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) criteria for major depressive disorder (recurrent and nonrecurrent course will be identified)
* Score of 16 or higher on the 24-item Hamilton Depression Rating Scale (HDRS) at study entry
* Score of 26 or higher on the Mini-Mental State Exam (MMSE)

Exclusion Criteria:

* History of psychiatric illness or a substance abuse disorder other than unipolar depression, diagnosed prior to the onset of the first depressive episode
* Presence of psychotic symptoms
* Severe or acute medical illness (e.g., major surgery, metastatic cancer, stroke, heart attack) 6 months prior to study entry
* Acute suicidal or violent behavior or history of suicide attempt within the year prior to study entry
* Presence of delirium, neurodegenerative dementia, Parkinson's disease, or any other central nervous system (CNS) diseases
* Toxic or metabolic abnormalities on laboratory examination
* Medications taken or medical illnesses present that could account for depression
* Active heart failure categorized as Class III or greater according to New York Heart Association criteria
* Heart attack or crescendo angina within the 3 months prior to study entry
* Symptomatic cardiac arrhythmias or symptomatic, hemodynamically significant mitral or aortic valvular disease
* Resting heart rate less than 50 beats per minute and a corrected QT (QTc) interval greater than 0.45 seconds
* Second or third degree atrioventricular block
* Systolic blood pressure greater than 180 mmHg or less than 90 mmHg and diastolic blood pressure greater than 105 mmHg or less than 50 mmHg at study entry
* Treated with depot neuroleptic therapy within 6 months prior to study entry
* Treated with any neuroleptic, antidepressant, anxiolytic medication (other than lorazepam), or over-the-counter CNS-active medications used for treatment of depression (e.g, St. John's Wort, kava-kava, melatonin) within 2 weeks (4 weeks for fluoxetine or monoamine-oxidase inhibitors (MAOIs)) prior to the first administration of study medication
* Known allergy to citalopram or MPH or history of ineffective treatment with citalopram or MPH for current depressive episode
* Requires concomitant therapy with any prescription or over-the-counter medications that have potentially dangerous interactions with either citalopram or MPH
* Requires electroconvulsive therapy (ECT) or received ECT within 3 months prior to study entry
* Initiated psychotherapy within 3 months prior to study entry or will be initiating or terminating psychotherapy during the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2008-02; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lavretsky, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute - Neuropsychiatric Institute (NPI), Los Angeles, California, United States

REFERENCES:
- [Result] Schneider B, Ercoli L, Siddarth P, Lavretsky H. Vascular burden and cognitive functioning in depressed older adults. Am J Geriatr Psychiatry. 2012 Aug;20(8):673-81. doi: 10.1097/JGP.0b013e31822ccd64. PMID 21857219
- [Derived] Eyre HA, Eskin A, Nelson SF, St Cyr NM, Siddarth P, Baune BT, Lavretsky H. Genomic predictors of remission to antidepressant treatment in geriatric depression using genome-wide expression analyses: a pilot study. Int J Geriatr Psychiatry. 2016 May;31(5):510-7. doi: 10.1002/gps.4356. Epub 2015 Oct 15. PMID 26471432

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 181 participants were enrolled in the study and 38 participants dropped out before randomization. A total of 143 participants were assigned to groups.
Groups:
- 1 - Citalopram + Placebo: Participants will take a combination of citalopram and placebo for 16 weeks
  Citalopram: Citalopram dosage will be 20 to 60 mg a day. Participants will begin taking one 20-mg capsule once per day, and this dosage may be increased or decreased depending on the participant's response to the medication. Participants will continue on their assigned dosage of citalopram until treatment completion.
  Placebo: Placebo pills will be taken in combination with the active pills. Participants will initially take 1 capsule twice per day, which will be increased to a maximum of 16 capsules twice per day. After Visit 11, placebo dosage will be gradually reduced over 2 weeks until participants are no longer taking any capsules.
- 2 - Methylphenidate + Placebo: Participants will take a combination of methylphenidate and placebo for 16 weeks
  Methylphenidate (MPH): MPH dosage will be 5 to 40 mg a day. Participants will initially take 1 capsule twice per day, which will be increased to a maximum of 16 capsules twice per day. After Visit 11, MPH dosage will be gradually reduced over 2 weeks until participants are no longer taking any capsules.
  Placebo: Placebo pills will be taken in combination with the active pills. Participants will initially take 1 capsule twice per day, which will be increased to a maximum of 16 capsules twice per day. After Visit 11, placebo dosage will be gradually reduced over 2 weeks until participants are no longer taking any capsules.
- 3 - Methylphenidate + Citalopram: Participants will take a combination of methylphenidate and citalopram for 16 weeks
  Methylphenidate (MPH): MPH dosage will be 5 to 40 mg a day. Participants will initially take 1 capsule twice per day, which will be increased to a maximum of 16 capsules twice per day. After Visit 11, MPH dosage will be gradually reduced over 2 weeks until participants are no longer taking any capsules.
  Citalopram: Citalopram dosage will be 20 to 60 mg a day. Participants will begin taking one 20-mg capsule once per day, and this dosage may be increased or decreased depending on the participant's response to the medication. Participants will continue on their assigned dosage of citalopram until treatment completion.
Period: Overall Study
Arm/Group | 1 - Citalopram + Placebo | 2 - Methylphenidate + Placebo | 3 - Methylphenidate + Citalopram
Started | 48 | 48 | 47
Completed | 46 | 46 | 46
Not Completed | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 - Citalopram + Placebo | 2 - Methylphenidate + Placebo | 3 - Methylphenidate + Citalopram | Total
Number analyzed (Participants) | 48 | 48 | 47 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (7.1) | 70.0 (7.1) | 68.9 (7.6) | 69.7 (7.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 17 | 8 | 38
  >=65 years | 35 | 31 | 39 | 105
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 19 | 78
  Male | 17 | 20 | 28 | 65
Region of Enrollment [Number; unit: participants]
  United States | 48 | 48 | 47 | 143

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HDRS) Maintained Scores at Week 16
Description: The Hamilton Depression Rating Scale (HDRS) is a 24-item depression scale and the total score is summed with a minimum score=0 and maximum score=76. There are no subscales and the higher values represent a worse outcome. Outcomes are measured and defined as follows: 1) Response will be defined as HDRS scores of 10 or less; 2) Sustained response will be defined as maintained response at week 16; 4) Remission will be defined as HDRS scores of 6 or less.
Time Frame: Maintained response measured at Week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 - Citalopram + Placebo | 2 - Methylphenidate + Placebo | 3 - Methylphenidate + Citalopram
Number analyzed (Participants) | 48 | 48 | 47
units on a scale | 18.3 (5.2) [0 to 76] | 18.7 (5.1) [0 to 76] | 19.8 (6.3) [0 to 76]

2. Secondary Outcome: Quality of Life Assessment
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) is a 16 item self-administered questionnaire that captures life satisfaction over the past week. Each question is rated on a 5 point scale from 1 (Very Poor) to 5 (Very Good). The total score is reported for items 1-14. The minimum raw score on the Q-LES-Q-SF is 14, and the maximum score is 70 with higher values representing a better outcome.
Time Frame: Measured at Baseline and Week 16
Population: The overall analyzed at baseline and week 16 differs due to participant drop out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 - Citalopram + Placebo | 2 - Methylphenidate + Placebo | 3 - Methylphenidate + Citalopram
Number analyzed (Participants) | 48 | 47 | 48
units on a scale
  Baseline | 45.50 (7.59) | 47.06 (8.43) | 47.52 (7.32)
  Week 16: number analyzed (Participants) | 31 | 35 | 34
  Week 16 | 54.45 (7.54) | 53.54 (13.11) | 57.79 (9.19)

ADVERSE EVENTS:
Arm/Group | 1 - Citalopram + Placebo | 2 - Methylphenidate + Placebo | 3 - Methylphenidate + Citalopram
Serious Adverse Events (participants affected / at risk) | 1/48 | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 3/48 | 9/48 | 4/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 - Citalopram + Placebo (N=48) | 2 - Methylphenidate + Placebo (N=48) | 3 - Methylphenidate + Citalopram (N=47)
death (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 - Citalopram + Placebo (N=48) | 2 - Methylphenidate + Placebo (N=48) | 3 - Methylphenidate + Citalopram (N=47)
Reduced salivation (Gastrointestinal disorders) | 3 | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No